CLINICAL TRIAL: NCT00894439
Title: A Randomized, Open-label, Single-dose, 3-period Crossover Study to Describe the Pharmacokinetic Parameters of BLI-489 and Piperacillin When Administered Simultaneously Compared to When Each is Administered Alone.
Brief Title: Study Evaluating BLI-489 and Piperacillin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3219K1-1002
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — BLI-489; Piperacillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: BLI-489/Piperacillin; Drug: BLI-489; Drug: Piperacillin

INTERVENTIONS:
Drug: BLI-489/Piperacillin
Drug: BLI-489
Drug: Piperacillin

SUMMARY:
The purpose of this study is to evaluate how BLI-489 and piperacillin interact when given together to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women of non-childbearing potential, aged 18 to 50 years of age inclusive at screening.
2. Body mass index (BMI) in the range of 18 to 32 kg/m2 and body weight greater than or equal to 50 kg.
3. Healthy as determined by the investigator on the basis of the screening evaluations.
4. Nonsmoker of smoker of fewer than 10 cigarettes per day as determined by history.

Exclusion Criteria:

1. Presence of history of any disorder that may prevent the successful completion of the study.
2. History of drug abuse within 1 year.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics as evaluated by drug concentrations in the blood and urine. | 10 days

SECONDARY OUTCOMES:
Safety as measured by the number of adverse events and serious adverse events. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States